CLINICAL TRIAL: NCT00538564
Title: Tadalafil for Treatment of Priapism in Men With Sickle Cell Anemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial closed just prior to study receiving Investigational Review Board approval
Sponsor: Johns Hopkins University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NA_00004434
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Sickle Cell Anemia; Priapism
Keywords: prolonged, painful erection; priapism; sickle cell anemia
MeSH Terms: conditions — Anemia, Sickle Cell; Priapism | interventions — Tadalafil; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tadalafil (Experimental): Participants assigned to this arm were given oral 10 mg tadalafil tablets to take 3 times a week for 16 weeks.
  Interventions: Drug: tadalafil
- Placebo (Placebo Comparator): Participants assigned to this arm were given a placebo pill 3 times a week for the first 8 weeks, and then Tadalafil 10 mg 3 times a week for weeks 9-16.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tadalafil — 10mg oral tablets taken 3 times a week for 2 months
  Other Names: Cialis
  Arms: Tadalafil
Drug: placebo — Placebo tablets taken orally 3 times a week for 2 months
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
This research is being done to compare the effect of tadalafil with placebo (an inactive substance that looks like the study drug, but should have no effect) on the frequency of recurrent priapism (prolonged erection, unassociated with sexual interest or desire) and the nature of sexual experiences in male patients with sickle cell disease.

DETAILED DESCRIPTION:
This study will investigate phosphodiesterase 5 (PDE 5) inhibitor therapy as a potential treatment for recurrent ischemic priapism. Enrolled participants will be randomized to receive oral 10 mg tadalafil tablets 3 times a week or receive matching placebo. Patients will be instructed to use the medication in the morning a few hours after awakening from night time sleep, and they will be instructed against engaging in any form of sexual activity or excitement within 8 hours of dosing. Treatment duration will be 2 months for each participant. After the 2 month period, participants on tadalafil and placebo will be offered tadalafil (same dosing regimen) for an additional 2 months.

The study duration will be 4 months.

Tests and procedures will include: consent; medical history; physical examination; clinical laboratory tests; completion of questionnaires; and medication dispensation.

ELIGIBILITY:
Inclusion Criteria:

* All men (18 years of age and older) with actively recurrent ischemic priapism, defined as multiple, self-limited erectile events (characteristically less than 3 hours in duration) occurring repeatedly at least twice a week in the absence of sexual interest or desire may be considered for enrollment
* Able to swallow whole tablets equivalent to capsule size 0
* Available for protocol-specified visits and procedures

Exclusion Criteria:

* History of refractory-type priapism
* History of drug or alcohol abuse
* Currently smokes or has a 20 pack-year history of cigarette smoking
* Take any medications called "nitrates"
* History of acute or chronic depression
* History of heart problems such as angina, heart failure, irregular heartbeats or myocardial infarction
* History of low blood pressure or high blood pressure that is not controlled
* History of diabetes, liver problems, or kidney problems
* A glomerular filtration rate of <50ml/min.
* History of retinitis pigmentosa or severe vision loss, including a condition called NAION
* History of stomach ulcers
* History of HIV, multiple myeloma, or leukemia
* History of Peyronie's disease
* History of spinal trauma or surgery to the brain or spinal cord
* Any contraindications to Cialis use
* Currently participating in another clinical investigation

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
change in recurrent priapism frequency | From baseline to 2 months post treatment
  A "Priapism sexual activity log" will be administered to participants. In the log, participants will be asked to quantify the number of priapic episodes they have experienced in the previous 2 weeks according to the following scale/tiers: 0 = no episodes, 1 = 1-2 episodes, 2 = 3-4 episodes, 3 = 5-8 episodes and 6 = greater than 20 episodes.
change of recurrent priapism frequency | From 2 months post treatment to 4 months post treatment
  A "Priapism sexual activity log" will be administered to participants. In the log, participants will be asked to quantify the number of priapic episodes they have experienced in the previous 2 weeks according to the following scale/tiers: 0 = no episodes, 1 = 1-2 episodes, 2 = 3-4 episodes, 3 = 5-8 episodes and 6 = greater than 20 episodes.

SECONDARY OUTCOMES:
change in nature of sexual experiences | baseline to 2 months post treatment
  The International Index of Erectile Function (IIEF) will be administered. This is a 15 item questionnaire . The questionnaire measures Erectile Function (scored from 0-30), Intercourse satisfaction (0-15), orgasmic function (0-10), Sexual Desire (2-10) and Overall satisfaction (2-10).
change in nature of sexual experiences | 2 month post treatment to 4 months post treatment
  The International Index of Erectile Function (IIEF) will be administered. This is a 15 item questionnaire . The questionnaire measures Erectile Function (scored from 0-30), Intercourse satisfaction (0-15), orgasmic function (0-10), Sexual Desire (2-10) and Overall satisfaction (2-10)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur L. Burnett, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Outpatient Center; Johns Hopkins Medical Institutions, Baltimore, Maryland, United States